CLINICAL TRIAL: NCT05061940
Title: Screening Protocol to Assess the Expression of Tumor Associated Antigens (TAAs), Human Papillomavirus (HPV-16) Antigens and Human Leucocyte Antigen (HLA) Sub-Types in Patients With Head and Neck, Cervical, Melanoma and Non-Small Cell Lung Cancers.
Brief Title: This SCR-103 Protocol Will Permit Sites to Proactively Assess TAA, HLA and HPV-16 Status in Patients With Selected Solid Tumors to Determine Suitability for Repertoire Immune Medicines Treatment Protocols.
Status: Terminated | Type: Observational
Why Stopped: Development program terminated
Sponsor: Repertoire Immune Medicines (Industry)
Responsible Party: Sponsor
Other Study IDs: SCR-103
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Cancer; Melanoma; HPV-Related Malignancy; HPV-Related Carcinoma; HPV-Related Cervical Carcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma; Lung Cancer, Nonsmall Cell; Melanoma (Skin)
Keywords: HPV-16 E6/E7; TT-101; PRIME-102; Metastatic; Solid Tumor
MeSH Terms: conditions — Head and Neck Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tumor Profiling — Testing TAA and HPV expression. HLA typing.

SUMMARY:
The purpose of this study is to obtain archived tumor tissue or pre-existing antigen expression data from patients with Head and Neck, Cervical, Melanoma and Non-Small Cell Lung Cancers to assess antigen expression and patient suitability for a Repertoire Immune Medicines Treatment Protocol.

DETAILED DESCRIPTION:
This screening study is intended for men and women at least 18 years of age who have selected advanced solid tumors. The study will assess the patient's selected tumor antigens and/or HPV-16 E6/E7 expression profiles. Human leukocyte antigen (HLA) subtype will also be assessed.

Based on the results, it will be determined if a patient is eligible to be considered for a Repertoire Immune Medicines sponsored clinical trial(s) testing of the safety and efficacy of a multi-antigen cytokine-enhanced T cell therapy. No treatment intervention will occur as part of this screening study.

Upon enrollment, patients will be required to provide archival tumor tissue and saliva samples. Based upon the results of these diagnostic analyses, if eligible, patients may be enrolled in an appropriate interventional clinical trial(s) at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent
* Age ≥ 18 years
* Histologically- or cytologically-confirmed, relapsed/refractory, and metastatic or locally advanced head and neck, cervical, melanoma or non-small cell lung cancers. Other solid tumor types may be analyzed at the discretion of the Sponsor
* Able to provide archived tumor tissue or have existing data on TAAs, HPV status or HLA sub-type
* Willing to provide a saliva sample

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for inclusion in this study must meet all of the following criteria:
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects with the expression of multiple tumor associated antigens and/or HPV-16 E6/E7. | 5 years
  To identify patients with Head and Neck, Cervical, Melanoma and Non-Small Cell Lung Cancer that could potentially be eligible for Repertoire Immune Medicines clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: David Spriggs, MD, Study Director — Repertoire Immune Medicines
Locations (3):
- United States (3):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Sarah Cannon Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No